CLINICAL TRIAL: NCT04703270
Title: Understanding COVID-19 Infection in Pregnant Women and Their Babies
Acronym: periCOVID
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.0276
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-08

CONDITIONS: Corona Virus Infection; Pregnancy Related; Neonatal Infection; Breastfeeding
MeSH Terms: conditions — Coronavirus Infections; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposed: Expectant mothers with a positive nasopharyngeal swab for SARS-CoV-2 at any point during pregnancy from 24 weeks gestation regardless of antibody status.
- Seropositive: Expectant mothers with a negative nasopharyngeal swab for SARS-CoV-2 at any point during pregnancy from 24 weeks gestation but positive IgM/IgG antibodies against SARS-CoV-2.
- Unexposed: Expectant mothers with a negative nasopharyngeal swab for SARS-CoV-2 at any point during pregnancy from 24 weeks gestation and negative IgM/IgG antibodies against SARS-CoV-2.

SUMMARY:
This national study will recruit expectant mothers with and without positive nasopharyngeal swabs for SARS-CoV-2, and aims to determine the seroepidemiology of SARS-CoV-2 amongst expectant mothers and their infants in the U.K.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Any woman pregnant in selected hospitals in England who has no signs or symptoms of COVID-19 disease during pregnancy and is rtPCR negative at delivery
* Any woman pregnant in any hospital in England who tests positive by rtPCR at any point during pregnancy from 24 weeks gestation onwards, regardless of signs and symptoms

Exclusion Criteria:

* If the pregnant woman is under 18 years in prison or unable to make an informed consent for other reasons (e.g. learning difficulties, language barriers)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pregnant women ≥ 24 weeks gestation in England.
Sampling Method: Non-Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants had their antibodies against SARS-CoV-2 tested prior to assignment of a group.
Groups:
- Unexposed: Expectant mothers with a negative nasopharyngeal swab for SARS-CoV-2 at any point during pregnancy from 24 weeks gestation.
- Vaccinated: Expectant mothers with a negative nasopharyngeal swab for SARS-CoV-2 at any point during pregnancy from 24 weeks gestation who received a vaccine against SARS-CoV-2 prior to delivery.
- Vaccinated and Exposed: Expectant mothers with a positive nasopharyngeal swab for SARS-CoV-2 at any point during pregnancy from 24 weeks gestation who also received a vaccine against SARS-CoV-2 prior to delivery.
Period: Overall Study
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Started | 173 | 627 | 43 | 38
Completed | 173 | 627 | 43 | 38
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed | Total
Number analyzed (Participants) | 173 | 627 | 43 | 38 | 881
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.0 [29.0 to 36.0] | 31.0 [27.0 to 35.0] | 34.0 [30.5 to 37.0] | 33.5 [31.3 to 36.8] | 32.0 [28.0 to 32.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 627 | 43 | 38 | 881
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 85 | 496 | 32 | 24 | 637
  Asian/Asian British | 9 | 54 | 8 | 4 | 75
  Black African/Caribbean/British | 4 | 20 | 0 | 0 | 24
  Other | 8 | 12 | 2 | 1 | 23
  Mixed/Multiple | 1 | 12 | 0 | 0 | 13
  Not Stated | 66 | 33 | 1 | 9 | 109

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations in Maternal Blood in Pregnant Women in England
Description: Antibody concentrations in maternal blood in pregnant women in England: ADCD-S values reported
Time Frame: Delivery
Measure: Geometric Mean (Inter-Quartile Range); unit: CAU/ml
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 173 | 627 | 43 | 38
CAU/ml | 37.2 [13.2 to 102.1] | 7.2 [5.0 to 5.0] | 80.3 [31.9 to 228.3] | 590.5 [308.7 to 1094.8]

2. Primary Outcome: Antibody Concentrations in Cord/Infant Blood at Delivery
Description: Cord blood was tested to determine infant antibody levels; where a cord blood sample was not available, a blood sample was taken from the infant instead. ADCD-S assay results are presented.
Time Frame: Delivery
Population: Number of participants analysed represents all those for whom a sample was received that was sufficient for analysis with the assay.
Measure: Geometric Mean (Inter-Quartile Range); unit: CAU/mL
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 139 | 489 | 32 | 27
CAU/mL | 35.9 [11.7 to 88.4] | 7.5 [5.0 to 5.0] | 83.9 [29.8 to 227.8] | 549.0 [323.9 to 1314.7]

3. Secondary Outcome: Number of Participants With Breastmilk Samples Positive for Antibodies Specific to SARS-CoV-2
Description: Number of participants with breastmilk samples positive for antibodies specific to SARS-CoV-2
Time Frame: At birth
Population: Most participants did not provide a breastmilk sample of sufficient quantity for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 0 | 1 | 29 | 1
Participants |  | 0 | 16 | 0

4. Secondary Outcome: Number of Mother-infant Pairs Who Are Both rtPCR Positive for SARS-CoV-2 in Blood at Delivery
Time Frame: Delivery
Population: No sufficient samples were received to enable rtPCR testing of mother and baby within a pair after sample testing for the primary outcome.
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Mother-infant Pairs Who Are Both rtPCR Positive for SARS-CoV-2 in Secretions at Delivery
Time Frame: Delivery
Population: All pairs for which a neonatal sample was received for the delivery timepoint were analysed. No delivery secretion samples were taken from neonates in the Unexposed group as per the study protocol.
Measure: Number; unit: Number of mother-infant pairs
Arm/Group | Exposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 116 | 2 | 18
Number of mother-infant pairs | 0 | 0 | 0

6. Secondary Outcome: Breastmilk Samples That Are rtPCR Positive
Time Frame: Delivery
Population: No samples were received which were sufficient to allow PCR testing after antibody testing.
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Placental Samples That Are rtPCR Positive
Time Frame: Delivery
Population: The population numbers reflect the samples received which were suitable for rtPCR testing. No placental samples were received from participants in the Unexposed or Vaccinated arms, so these were not analysed.
Measure: Number; unit: No. of Placental Samples rtPCR positive
Arm/Group | Exposed | Vaccinated and Exposed
Number analyzed (Participants) | 109 | 15
No. of Placental Samples rtPCR positive | 1 | 0

8. Secondary Outcome: Number of Participants in Whose Placental Sample the Virus Can be Grown in Vitro
Time Frame: Delivery
Population: All PCR placental samples were negative at delivery, except for one swab which was determined to have likely been contaminated in the delivery room. As all other samples were negative, none proceeded to in vitro culture.
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants in Whose Breast Milk Sample the Virus Can be Grown in Vitro
Time Frame: Delivery
Population: No breastmilk samples were PCR positive, therefore none proceeded to in vitro culture.
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Mother-baby Pairs in Whom the Virus Can be Grown in Vitro
Time Frame: 6 weeks post delivery
Population: No paired samples proceeded to in vitro culture due to lack of PCR positivity.
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Over the study period, i.e. until 6 weeks postpartum.
Arm/Group | Exposed | Unexposed | Vaccinated | Vaccinated and Exposed
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/627 | 0/43 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/627 | 0/43 | 0/38
Other Adverse Events (participants affected / at risk) | 0/173 | 0/627 | 0/43 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04703270/Prot_SAP_000.pdf